CLINICAL TRIAL: NCT00599937
Title: Assessment of the Optimal Timing of Chemotherapy With or After ATRA and the Role of Maintenance
Brief Title: APL93: Timing of CxT and Role of Maintenance
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Groupe d'etude et de travail sur les leucemies aigues promyelocytaires (Other)
Collaborators: DRC lille, France (Unknown)
Responsible Party: DRC Lille, CHU Lille
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APL93
Record Dates: First submitted 2007-12-27; First posted 2008-01-24 (Estimated); Last update posted 2008-01-24 (Estimated); Status verified 2007-12

CONDITIONS: Leukemia, Promyelocytic, Acute
Keywords: APL
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute | interventions — Tretinoin; Maintenance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- ATRA ->Chemo (No Intervention): Patients 65 years of age with a WBC count less than 5,000 were randomized to receive the reference ATRA treatment of our previous trial (APL91 trial), ie, 45 mg/m2/d ATRA followed by CT or ATRA plus CT (ATRA+CT). In the ATRA followed byCT group, patients received 45 mg/m2/d ATRA orally until CR, with a maximum of 90 days. After CR achievement, they received a course of 60 mg/m2/d daunorubicin (DNR) for 3 days and 200 mg/m2/d AraC for 7 days (course I). However, course I was added to ATRA if the WBC count was increased to greater than 6,000, 10,000, or 15,000 by day 5, 10, and 15 of ATRA treatment, respectively, because, from our experience, patients were at risk of ATRA syndrome above those thresholds.
- ATRA+CT (Experimental): Patients randomized to the ATRA+CT group received the same combination of ATRA and CT, with course I of CT starting on day 3 of ATRA treatment. This 48-hour interval before onset of CT was based on our previous report, because it allowed correction of coagulopathy.
  Interventions: Drug: ATRA
- High WBC (No Intervention): Patients with a WBC count greater than 5,000 at presentation (irrespective of their age) and patients 66 to 75 years of age with a WBC count 5,000 were not randomized but received ATRA plus CT course I from day 1 (high WBC group) and the same schedule as in the ATRA->CT group (elderly group), respectively.
- no maintenance (No Intervention): No maintenance
- maintenance ATRA (Experimental): Intermitent ATRA as maintenance
  Interventions: Drug: ATRA and or Chemo as maintenance
- maintenance Cxt (Experimental): continuous CT with 6 mercaptopurine (90 mg/m2/d, orally) and methotrexate (15 mg/m2/wk, orally) as maintenance
  Interventions: Drug: ATRA and or Chemo as maintenance
- maintenance both (Experimental): continuous CT with 6 mercaptopurine (90 mg/m2/d, orally) and methotrexate (15 mg/m2/wk, orally) AND ATRA as maintenance
  Interventions: Drug: ATRA and or Chemo as maintenance

INTERVENTIONS:
Drug: ATRA — early introduction of ATRA
  Arms: ATRA+CT
Drug: ATRA and or Chemo as maintenance — patients were randomized both to receive or not receive intermittent ATRA (45 mg/m2/d, 15 days every 3 months) and to receive or not receive continuous CT with 6 mercaptopurine (90 mg/m2/d, orally) and methotrexate (15 mg/m2/wk, orally), according to a 2-by-2 factorial design stratified on the initial induction treatment group
  Other Names: ATRA
  Arms: maintenance ATRA; maintenance Cxt; maintenance both

SUMMARY:
Objectives of the trial were to assess the optimal timing of chemotherapy with or after ATRA and the role of maintenance therapy.

DETAILED DESCRIPTION:
Induction treatment was stratified by age and initial WBC count. Patients ≤65 years of age with a WBC count less than 5,000/µL were randomized to receive the reference ATRA treatment of our previous trial (APL91 trial) {Fenaux, 1993 #2088}, ie, 45 mg/m2/d ATRA followed by CT (ATRA→CT group) or ATRA plus CT (ATRA+CT). In the ATRA→CT group, patients received 45 mg/m2/d ATRA orally until CR, with a maximum of 90 days. After CR achievement, they received a course of 60 mg/m2/d daunorubicin (DNR) for 3 days and 200 mg/m2/d AraC for 7 days (course I). However, course I was added to ATRA if the WBC count was increased to greater than 6,000/µL, 10,000/µL, or 15,000/µL by day 5, 10, and 15 of ATRA treatment, respectively, be-cause, from our experience, patients were at risk of ATRA syndrome above those thresholds{de Botton, 2003 #1127; De Botton, 1998 #1604}. Patients randomized to the ATRA+CT group received the same combination of ATRA and CT, with course I of CT starting on day 3 of ATRA treatment.

Patients with a WBC count greater than 5,000/µL at presentation (irrespective of their age) and patients 66 to 75 years of age with a WBC count ≤ 5,000/µL were not ran-domized but received ATRA plus CT course I from day 1 (high WBC group) and the same schedule as in the ATRA→CT group (elderly group), respectively.

Treatment of coagulopathy during the induction phase was based on platelet support to maintain the platelet count at a level greater than 50,000 /µL until the disappea-rance of coagulopathy. The use of heparin, tranexamic acid, fresh frozen plasma, and fibrinogen transfusions was optional.

CR patients received 2 CT consolidation courses, including course II (identical to course I) and course III, consisting of 45 mg/m2/d DNR for 3 days and 1 g/m2 AraC every 12 hours for 4 days. The elderly group only received course II.

Three to 4 weeks after hematological recovery from this consolidation CT, patients who were still in CR were randomized both to receive or not receive intermittent ATRA (45 mg/m2/d, 15 days every 3 months) and to receive or not receive continuous CT with 6 mercaptopurine (90 mg/m2/d, orally) and methotrexate (15 mg/m2/wk, oral-ly), according to a 2-by-2 factorial design stratified on the initial induction treatment group. Maintenance treatment was scheduled for 2 years. Randomizations for induc-tion and maintenance, stratified on center, were performed through a centralized tele-phone assignment procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of APL, based on morphology criteria
2. Age 75 years or less; and
3. Written informed consent. Diagnosis had to be subsequently confirmed by presence of t(15;17) or PML-RAR gene rearrangement. In the absence of t(15;17) and if no analysis of the rearrangement could be made, review of initial marrow slides by an independent morphologist was mandatory.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 576 (Actual)
Dates: Start 1993-01; Primary Completion 1998-12 (Actual); Study Completion 1998-12 (Actual)

PRIMARY OUTCOMES:
For induction treatment event-free survival (EFS), calculated from the date of randomization, was the major endpoint. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: pierre fenaux, mD, Principal Investigator — Assistance Publique Hopitaux de Paris

REFERENCES:
- [Result] Fenaux P, Chastang C, Chevret S, Sanz M, Dombret H, Archimbaud E, Fey M, Rayon C, Huguet F, Sotto JJ, Gardin C, Makhoul PC, Travade P, Solary E, Fegueux N, Bordessoule D, Miguel JS, Link H, Desablens B, Stamatoullas A, Deconinck E, Maloisel F, Castaigne S, Preudhomme C, Degos L. A randomized comparison of all transretinoic acid (ATRA) followed by chemotherapy and ATRA plus chemotherapy and the role of maintenance therapy in newly diagnosed acute promyelocytic leukemia. The European APL Group. Blood. 1999 Aug 15;94(4):1192-200. PMID 10438706
- [Derived] Ades L, Guerci A, Raffoux E, Sanz M, Chevallier P, Lapusan S, Recher C, Thomas X, Rayon C, Castaigne S, Tournilhac O, de Botton S, Ifrah N, Cahn JY, Solary E, Gardin C, Fegeux N, Bordessoule D, Ferrant A, Meyer-Monard S, Vey N, Dombret H, Degos L, Chevret S, Fenaux P; European APL Group. Very long-term outcome of acute promyelocytic leukemia after treatment with all-trans retinoic acid and chemotherapy: the European APL Group experience. Blood. 2010 Mar 4;115(9):1690-6. doi: 10.1182/blood-2009-07-233387. Epub 2009 Dec 17. PMID 20018913